CLINICAL TRIAL: NCT00397176
Title: Ascending, Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of DVS SR Administered Orally to Healthy Japanese Female Subjects
Brief Title: Study Evaluating Safety, Tolerability, and PK of DVS SR in Healthy Japanese Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 3151A2-1200
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Vasomotor Symptoms

INTERVENTIONS:
Drug: desvenlafaxine succinate sustained release (DVS SR)

SUMMARY:
Safety, tolerability, and pharmacokinetics (PK) of desvenlafaxine succinate sustained release (DVS SR) in healthy Japanese female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, first-generation (born in Japan, living in the US for less than 5 years)
* Japanese female subjects

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2006-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Safety, Tolerability, PK

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer